CLINICAL TRIAL: NCT02145104
Title: Comparison of the Efficacy and Safety of Cilnidipine 10mg/Valsartan 160mg Combination Therapy, Cilnidipine 5mg/Valsartan 160mg Combination Therapy and Valsartan 160mg Monotherapy in Hypertensive Patients Inadequately Controlled With Valsartan 160mg Monotherapy: a Multicenter, Randomized, Double Blind Phase III Study
Brief Title: Efficacy/Safety of Cilnidipine Plus Valsartan Versus Valsartan in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID_IDCV_1302
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; cilnidipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): cilinidpine 10mg + valsartan 160mg
  Interventions: Drug: valsartan 160mg, cilnidipine 10mg, cilinidipine 5mg
- Arm B (Experimental): cilnidipine 5mg + valsartan 160mg
  Interventions: Drug: valsartan 160mg, cilnidipine 10mg, cilinidipine 5mg
- Arm C (Active Comparator): valsartan 160mg
  Interventions: Drug: valsartan 160mg, cilnidipine 10mg, cilinidipine 5mg

INTERVENTIONS:
Drug: valsartan 160mg, cilnidipine 10mg, cilinidipine 5mg

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of cilinidipine plus valsartan and valsartan alone in patients with essential hypertension inadequately controlled on valsartan monotherapy

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension patients whose blood pressure is not controlled before the study (sDBP≥90mmHg for drug-treated patients, sDBP≥95mmHg for drug-naive patients)

Exclusion Criteria:

* sSBP≥80mmHg after 4weeks of valsartan 160mg treatment
* has a history of hypersensitivity to dihydropyridines or angiotensin II receptor blockers

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
change from baseline in mean sDBP | 8 weeks

SECONDARY OUTCOMES:
change from baseline in mean sDBP | 4 weeks
change from baseline in mean sSBP | 4, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ju Choi, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyung-gi, South Korea